CLINICAL TRIAL: NCT03720262
Title: Prevention of Hernia After Loop Ileostomy Reversal
Acronym: PHaLIR
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Stockholm South General Hospital (Other)
Responsible Party: Principal Investigator, Åsa Hallqvist Everhov, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHaLIR
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Loop Ileostomy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the surgeon performing the follow-up are masked for the allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mesh reinforcement (Experimental): Retro muscular mesh at the stoma site.
  Interventions: Combination Product: Mesh reinforcement
- No reinforcement (Placebo Comparator): Standard closure of the abdominal wall
  Interventions: Other: No reinforcement

INTERVENTIONS:
Combination Product: Mesh reinforcement — Reinforcement of the abdominal wall with Ultrapro Advanced.
  Arms: Mesh reinforcement
Other: No reinforcement — Suturing the abdominal wall without mesh reinforcement
  Arms: No reinforcement

SUMMARY:
PHaLIR is a prospective, double-blinded randomized study in which patients planned for stoma reversal after rectal cancer surgery are randomized between retro muscular mesh Ultrapro Advanced or standard treatment without mesh.

DETAILED DESCRIPTION:
A temporary loop ileostomy is widely used when operating rectal cancer. The ostomy is then reversed in a separate operation. Morbidity of stoma reversal is significant, but not clearly defined. One complication in connection with stoma closure is development of hernia at the former stoma site.

A hernia is a weakening of the muscular layers and the connective tissue of the abdominal wall, which may cause pain and discomfort, as well as an inconvenient bulge. A hernia could also cause more serious complication of obstructed or strangulated bowel. According to international studies, the incidence of hernia at the ostomy site varies between 7% and 35%. Many of the studies are heterogenic and some of them include both colostomies and ileostomies. Among studies that focus on reversal of ileotomies the hernia incidence varies between 11-15%. Preliminary results from a retrospective study in Stockholm indicates a frequency of 7,9%.

The best method to avoid hernia after stoma closure is not known. Most commonly surgeons tend to close the fascia in one layer with monofilament suture. In the study mentioned above 91% of the operations were done with one-layer monofilament, mostly PDS. Use of prophylactic mesh in the abdominal wall has been proposed, but there is currently insufficient scientific evidence to recommend it as a routine.

The present study is focused on loop ileostomy closure after rectal cancer. A non-heterogenous group of ostomies will serve as a base to evaluate whether the incidence of hernia may be reduced. If this study detects a decreased frequency of hernia when using prophylactic meshes, it may lead to new recommendations for this patient group.

PHaLIR is a prospective, double-blinded randomized study in which patients planned for stoma reversal after rectal cancer surgery will be randomized to retro muscular mesh Ultrapro Advanced or standard treatment without mesh. Operating time, complications, LOS, pain, infections and postoperative hernia are to be studied. The patients will be identified and asked about participation when they come for postoperative control after rectal cancer operation and are planned for the ileostomy reversal after check of the rectal anastomosis. They will be given oral and written information and signed informed consent is required from all patients.

At operation the operation-protocol should be filled in. The operation notes will be written in a blinded way and the original version will be stored on paper until after the study is finished and then added to the patient chart.

At discharge from the surgical ward the patient should be planned for a follow up at the surgical clinic at 30 days postoperatively. The doctor at the follow up visit should be another than the operating surgeon. The patients should then fill in a questionnaire and the surgeon should note the postoperative complications in the 30-days follow up form. At the 30-day follow up the surgeon checks that the one-year follow up after the cancer operation is commissioned. Normally this is a CT thorax and abdomen with contrast. For the study-patients it should be complemented with the question of hernia and the CT scan shall be a CT with straining. The normal 1-year follow up for the cancer will be the follow up for the ileostomy reversal also. That means that in most cases it will take place 6-9 months after the reversal. At this control and at the three years control (after cancer operation) the patient will be given or mailed a questionnaire (the same as the 30-day questionnaire). The follow up by doctor could be done either with a clinical visit or a telephone call according to the routines of the clinic when they follow up their cancer patients. At three years follow up after cancer operation patients will also get the same questionnaire and the CT scan follow up at three years will also be with straining.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated for low anterior resection for rectal cancer with a diverting loop ileostomy and planned for stoma reversal

Exclusion Criteria:

* Language barrier or cognitive disability
* Recurrent cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Hernia | One year
  Hernia at the site of the stomal closure

SECONDARY OUTCOMES:
Operation time | Three hours
  Total operation time
Time for closing the stoma site | One hour
  Time required to close the stoma site
Hospital stay | Seven days
  Days to discharge
Postoperative pain | Thirty days
  Pain assessed on a Visual analogue scale ranging from 0 to 100, without subscales. 0 corresponds to no pain and 100 the most intense pain sensation imaginable.
Postoperative complications | Thirty days
  Complications, including surgical site infections

CONTACTS AND LOCATIONS:
Overall Officials: Åsa Hallqvist Everhov, MS, PhD, Principal Investigator — Stockholm South General Hospital
Locations (4):
- Sweden (4):
  - Södertälje Hospital, Södertälje
  - Stockholm South General Hospital, Stockholm
  - Ersta Hospital, Stockholm
  - Västmanland Hospital, Västerås

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eklov K, Bringman S, Lofgren J, Nygren J, Everhov AH. PHaLIR: prevent hernia after loop ileostomy reversal-a study protocol for a randomized controlled multicenter study. Trials. 2023 Sep 8;24(1):575. doi: 10.1186/s13063-023-07430-w. PMID 37684648